CLINICAL TRIAL: NCT01521429
Title: Longitudinal Study of Bone and Endocrine Disease in Children with MPS I, II, and VI: a Multicenter Study of the Lysosomal Disease Network.
Brief Title: Longitudinal Study of Bone Disease in Children with Mucopolysaccharidoses (MPS) I, II, and VI
Status: Completed | Type: Observational
Sponsor: Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center (Other)
Collaborators: Rare Diseases Clinical Research Network (Network); National Institute of Neurological Disorders and Stroke (NINDS) (NIH); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); UCSF Benioff Children's Hospital Oakland (Other); National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Principal Investigator, Lynda E Polgreen, Assistant Professor, Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center
Other Study IDs: 0906M68810; U54NS065768 (NIH)
Record Dates: First submitted 2011-11-11; First posted 2012-01-30 (Estimated); Last update posted 2024-10-22 (Actual); Status verified 2019-11

CONDITIONS: Mucopolysaccharidoses
MeSH Terms: conditions — Mucopolysaccharidoses

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum, plasma, white cells for DNA extraction, and urine will be retained.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- MPS I: Mucopolysaccharidosis I (Hurler, Scheie, Hurler-Scheie)
- MPS II: Mucopolysaccharidosis II (Hunter)
- MPS VI: Mucopolysaccharidosis VI (Maroteaux-Lamy)

SUMMARY:
Approximately 85% of individuals with Mucopolysaccharidosis (MPS) type I, II, or VI report weekly pain and 50-60% have significant limitations in their activities of daily living due to MPS related musculoskeletal disease despite treatment with enzyme replacement therapy (ERT). Thus there is a critical need to identify additional therapies to alleviate the burden of musculoskeletal disease in order to improve the health and quality of life of individuals with MPS. However, disease progression needs to be quantified to be able to determine efficacy of new therapies. This study is a multi-institutional, 5-year, longitudinal study of musculoskeletal disease in MPS. The objective is to quantitatively describe the progression of skeletal disease and identify biomarkers that either predict disease severity or could be used as therapeutic targets in individuals with MPS I, II, and VI. A database of standardized measurements of musculoskeletal disease in MPS will allow the field to efficiently move forward with therapeutic clinical trials in patients with MPS.

DETAILED DESCRIPTION:
Although children with MPS I, II, and VI who are treated with hematopoietic cell transplantation (HCT) and/or enzyme replacement therapy (ERT) are now living into adulthood with good cognitive development, their quality of life is significantly impacted by their skeletal abnormalities (i.e., kyphosis, scoliosis, genu valgum), joint contractures, pain, and severe short stature. Additional therapies (e.g., post-HCT supplemental ERT, anti-TNFα drugs, stop codon suppression drugs, gene therapy) to decrease the burden of skeletal disease and improve growth are needed. However, prior to these therapeutic studies, control data quantifying the progression of skeletal disease in individuals with MPS I, II and VI treated with ERT and/or HCT are needed, along with biomarkers to be used as early predictors of response to treatment.

Osteoporosis has been described in animal models of MPS. It is unknown whether abnormalities seen in animal models of MPS can be extrapolated to osteoporosis or increased risk of fracture in children and adults affected with MPS. Preliminary data suggest that children and adolescents with MPS I, II and VI have low bone mineral density (BMD) after adjustment for short stature and abnormal bone geometry and that markers of bone remodeling are cross-sectionally associated with BMD. It is unknown whether this decreased BMD during childhood will result in osteoporosis and increased fracture risk in adulthood. Determining the risk for osteoporosis in MPS I, II and VI has become particularly important as these individuals are now healthier and more mobile with new and improved treatments and thus have a greater opportunity for fracture.

Glycosaminoglycan (GAG) deposition has been identified in bone and cartilage in animal models of MPS. GAG deposition in cartilage has specifically been shown to induce inflammation (e.g. increased tumor necrosis-alpha [TNF- α ] levels in serum and synovial fluid), chondrocyte apoptosis, and hyperplasia of the synovial membranes. We have found that serum TNF-α is elevated in children and adolescents with MPS I, II and VI and is associated with bodily pain and poor physical function.

Our long-term goal is to identify and test new therapies for musculoskeletal disease in MPS. The objective of this proposed longitudinal observational study is to document the progression of skeletal disease and identify biomarkers that either predict disease severity or could be used as therapeutic targets in individuals with MPS I, II, and VI. The rationale for this project is to obtain baseline data for future therapeutic clinical trials and to identify potential therapeutic targets. Our central hypothesis is that skeletal disease will progress over time and that biomarkers of inflammation, and bone and cartilage turnover, will predict the severity of skeletal disease over time. Therefore, this study has the following specific aims (SA):

SA1: To characterize the progression of skeletal disease from childhood into young adulthood for individuals with MPS I, II and VI. Our hypothesis is that there will be a progressive decrease in bone health as this population matures into young adulthood due to decreasing mobility, chronic inflammation, and intrinsic MPS related bone disease.

SA2: To identify prognostic biomarkers of inflammation, bone remodeling, and cartilage turnover that can predict the progression of skeletal disease and impaired physical function in MPS I, II and VI. Our hypothesis is that biomarkers of inflammation, bone remodeling, and cartilage turnover, will be predictive of change in physical function, BMD, range of motion, hip dysplasia, kyphoscoliosis, quality of life, and height over 5 years.

At the completion of this study we expect to quantify the progression of skeletal disease in MPS I, II and VI treated with ERT and/or HCT to be used in future therapeutic clinical trials. In addition, we will obtain biomarkers of skeletal disease progression that could identify early treatment efficacy. Finally, we will gain further insight into the mechanism of persistent skeletal disease in MPS that will provide potential therapeutic targets.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of MPS I, II, or VI
* Ability to travel to study center for evaluations.
* Age ≥ 5 years and < 35 years: age at entry into study must be ≥5 years and ≤33 years to ensure a minimum of 2 study visits.

Exclusion Criteria:

* Pregnancy (will be determined at each study visit)
* Participation in any other study within the past 12 months which would result in increasing the child's radiation exposure above 500 mrem for the calendar year.
* Participants who cannot comply with study procedures or have other factors that would inhibit their participation as determined by the PI's discretion.

Ages: 5 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: community sample
Sampling Method: Non-Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2009-08; Primary Completion 2019-07-31 (Actual); Study Completion 2019-07-31 (Actual)

PRIMARY OUTCOMES:
Annual change in dual energy x-ray absorptiometry (DXA) | baseline, year 1, year 2, year 3
  Measurement of bone density and body composition

SECONDARY OUTCOMES:
Annual change in Peripheral quantitative computer tomography (pQCT) | baseline, year 1, year 2, year 3
  Measurement of volumetric bone density, bone geometry, bone strength, and muscle fat
Annual change in Biomarkers of bone remodeling | baseline, year 1, year 2, year 3
  Measurements of bone turnover
Annual change in Biodex | baseline, year 1, year 2, year 3
  Measurement of muscle strength
Annual change in Endocrine function tests | baseline, year 1, year 2, year 3
  Thyroid function, growth factor levels, pubertal hormones, vitamin D
Annual change in growth measurements | baseline, year 1, year 2, year 3
  sitting and standing heights, arm and tibial length

CONTACTS AND LOCATIONS:
Overall Officials: Lynda E Polgreen, MD, MS, Principal Investigator — Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center
Locations (3):
- United States (3):
  - Children's Hospital & Research Center Oakland, Oakland, California
  - Los Angeles Biomedical Research Institute at Harbor-UCLA Medical Center, Torrance, California
  - University of Minnesota, Minneapolis, Minnesota